CLINICAL TRIAL: NCT02199106
Title: Effectiveness of Neuronavigated Continuous Theta Burst Stimulation of the Left Heschl's Gyrus in Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Collaborators: University of Wuerzburg (Other); University Hospital Tuebingen (Other); University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, PhD, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ti-cTBS
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left temporal verum cTBS (Experimental): Continuous theta burst stimulation (MC-B70, MagPro,MagOption, Medtronic, Germany): 400 triplets of stimuli (triplets with 50Hz) at an frequency of 5Hz (in sum 1200 stimuli) with a break after 200 bursts over the left Heschl's gyrus targeted with anatomical neuronavigation (Localite, Germany); 30% maximum stimulator output (each session)
  Intervention: Left temporal verum cTBS
  Interventions: Device: Left temporal verum cTBS
- Left temporal placebo cTBS (Experimental): Continuous theta burst stimulation (MC-B70, MagPro,MagOption, Medtronic, Germany): 400 triplets of stimuli (triplets with 50Hz) at an frequency of 5Hz (in sum 1200 stimuli) with a break after 200 bursts over the left Heschl's gyrus targeted with anatomical neuronavigation (Localite, Germany); 30% maximum stimulator output (each session); coil tilted by 45° over both wings
  Intervention: Left temporal placebo cTBS
  Interventions: Device: Left temporal placebo cTBS

INTERVENTIONS:
Device: Left temporal verum cTBS — Continuous theta burst stimulation (MC-B70, MagPro,MagOption, Medtronic, Germany): 400 triplets of stimuli (triplets with 50Hz) at an frequency of 5Hz (in sum 1200 stimuli) with a break after 200 bursts over the left Heschl's gyrus targeted with anatomical neuronavigation (Localite, Germany); 30% maximum stimulator output (each session)
  Arms: Left temporal verum cTBS
  Other Names: MC-B70, MagPro,MagOption, Medtronic, Germany
  Arms: Left temporal verum cTBS
Device: Left temporal placebo cTBS — Continuous theta burst stimulation (MC-B70, MagPro,MagOption, Medtronic, Germany): 400 triplets of stimuli (triplets with 50Hz) at an frequency of 5Hz (in sum 1200 stimuli) with a break after 200 bursts over the left Heschl's gyrus targeted with anatomical neuronavigation (Localite, Germany); 30% maximum stimulator output (each session); coil tilted by 45° over both wings
  Arms: Left temporal placebo cTBS
  Other Names: MC-B70, MagPro,MagOption, Medtronic, Germany
  Arms: Left temporal placebo cTBS

SUMMARY:
Neuronavigated continuous theta burst stimulation of the left Heschl's gyrus is used to modulate auditory cortex activity and plasticity contributing to the perception and distress of chronic tinnitus.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. One significant modulator of tinnitus is stress. Tinnitus has been shown to be generated in the brain, as a result of functional reorganization of auditory neural pathways and the central auditory system. Repetitive transcranial magnetic stimulation (rTMS) is also effective in treatment of tinnitus with moderate effect size. Pilot data were positive for low-frequency rTMS applied to the temporal and temporoparietal areas. Continuous theta burst stimulation (cTBS) is a new protocol of rTMS with a possible superior effect in contrast to low-frequency rTMS. Also anatomical neuronavigation might increase the efficacy of rTMS due to exact targeting of the primary auditory cortex. Thus, the aim of this study is the evaluation of the clinical efficacy of neuronavigated left-sided cTBS in chronic tinnitus in a randomised sham-controlled two-arm design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bothersome, subjective chronic tinnitus
* Duration of tinnitus more than 6 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* acute or chronic inflammation of the middle ear, Meniere diseases, sudden idiopathic hearing loss, fluctuating hearing
* history of seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Change in tinnitus questionnaire total score (contrast baseline (-day 3) versus end of treatment (day 10)) | -day 3; day 10

SECONDARY OUTCOMES:
Change of tinnitus questionaire total score (all baseline (-week 2, - week1, - day 3) vs. all follow-up visits (day 6, day 10, week 1, week 3, week 8)) | -week 2; - week1; - day 3; day 6; day 10; week 1; week 3; week 8
Change of tinnitus handicap inventory total score (all baseline (-week 2, - week1, - day 3) vs. all follow-up visits (day 6, day 10, week 1, week 3, week 8)) | -week 2; - week1; - day 3; day 6; day 10; week 1; week 3; week 8
Change of tinnitus numeric rating scales (all baseline (-week 2, - week1, - day 3) vs. all follow-up visits (day 6, day 10, week 1, week 3, week 8)) | -week 2; - week1; - day 3; day 6; day 10; week 1; week 3; week 8
Change of depressive symptoms as measured by the Beck Depression Inventory II (BDI) (baseline visit -week 2 vs. all follow-up visits (day 6, day 10, week 1, week 3, week 8)) | -week 2; day 6; day 10; week 1; week 3; week 8

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Principal Investigator — University of Regensburg
Locations (4):
- Germany (4):
  - University of Muenster, Münster
  - University of Regensburg - Dept of Psychiatry, Regensburg
  - University of Tuebingen, Tübingen
  - University of Wuerzburg, Würzburg